CLINICAL TRIAL: NCT01702168
Title: Implementation of Cognitive Processing Therapy (CPT) for Posttraumatic Stress Disorder (PTSD) in Diverse Communities
Brief Title: Implementation of CPT for PTSD in Diverse Communities
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Luana Marques, Assistant in Psychology, Massachusetts General Hospital
Other Study IDs: 1K23MH096029-01A1 (NIH)
Record Dates: First submitted 2012-10-03; First posted 2012-10-05 (Estimated); Last update posted 2019-03-08 (Actual); Status verified 2019-03

CONDITIONS: Stress Disorders, Post-Traumatic
Keywords: PTSD; EBT; EST; Community; Latino
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- CBT Training
  Interventions: Other: Provider training: Cognitive Processing Therapy (CPT)

INTERVENTIONS:
Other: Provider training: Cognitive Processing Therapy (CPT)

SUMMARY:
Aim: To identify, assess, and address organizational context and provider-level barriers and facilitators of implementation of Evidence-based treatments (EBTs) using a mixed-methods approach in a diverse community mental health center (CMHC), Massachusetts General Hospital Chelsea Health Clinic (MGH Chelsea).

Hypothesis: Anticipated barriers may include, but are not limited to, organizational climate, heavy case-loads, community mental health workers (CMHW) beliefs about EBTs, and provider motivation to learn EBT.

ELIGIBILITY:
Inclusion Criteria:

* Be over 18 years of age
* Speak English
* Be employed at least part time at MGH
* Willing to have focus group/interview audiotaped and transcribed for data analysis

Exclusion Criteria:

* inability to meet the above inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We will be working with community mental health workers and stakeholders at a community clinic, MGH Chelsea.
Sampling Method: Non-Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2012-10; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
EBPAS-50 | up to 5 years
  Evidence Based Practice Attitudes Scale (EBPAS-50) is a brief, validated measure of clinician attitudes towards evidence based treatments (EBTs) containing four subscales: 1) Appeal measures whether the provider would adopt a new practice if it is intuitively appealing, or is being used by colleagues who are happy with it; 2)Requirement measures whether provider would adopt a practice if it is required by an agency, supervisor, or state; 3)Openness measures whether the provider is generally open to trying new interventions and would be willing to try or use new types of therapy, and 4)Divergence measures whether the provider perceives research-based interventions as not clinically useful or less important than clinical experience.
ORC | up to 5 years
  Organizational Readiness for Change (ORC) measures organizational climate. The ORC is defined as the organizational and staff factors related to adoption of new technologies. ORC is conceptualized as a set of factors that are necessary for sustained change. These factors include motivation, resources, staff attributes, and organizational climate. Readiness for change has been associated with successful dissemination.
OSC | up to 5 years
  The Organizational Social Context (OSC) measures the following domains: structure, culture, psychological and organizational climate, and work attitudes. The OSC measurement system is a validated measure guided by a model of social context that composes both organizational(structure and culture) and individual (work attitudes and behavior) level constructs, including individual and shared perceptions (psychological and organizational climate) that are believed to mediate the impact of the organization on the individual. The OSC measurement system includes 105 items that form 16 first order factors and seven second order factors confirmed in national samples of social and mental health service organizations. These factors are grouped by the domains of structure, culture, psychological and organizational climate, and work attitudes.

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital Chelsea Health Center, Chelsea, Massachusetts, United States